CLINICAL TRIAL: NCT02920307
Title: Prospective, Randomized and Controlled Study Comparing Fixation Versus no Fixation of Mesh in Laparoscopic Inguinal Hernia Repair
Brief Title: Study of Laparoscopic Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Park Gaziantep Hospital (Other)
Collaborators: Muğla Sıtkı Koçman University (Other); Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, Principal Investigator, Medical Park Gaziantep Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MK-002-LHR
Record Dates: First submitted 2016-09-22; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Hernia, Inguinal; Inguinal Hernia, Direct; Inguinal Hernia, Indirect; Hernia, Femoral; Recurrence; Neuralgia, Atypical; Neuralgia, Ilioinguinal; Neuralgia, Iliohypogastric Nerve
Keywords: laparoscopic inguinal hernia repair; total extraperitoneoscopic hernia repair; transabdominal preperitoneal hernia repair; inguinal hernia; laparoscopy; hernia repair; herniorraphy; laparoscopic surgery
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Recurrence; Neuralgia | interventions — tetraethylpyrazine; tetra-4-amidinophenoxypropane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TEP without fixation (Experimental): Standard totally extraperitoneoscopic preperitoneal (TEP) hernia repair without mesh fixation
  Interventions: Procedure: TEP without fixation
- TEP with fixation (Active Comparator): Standard totally extraperitoneoscopic preperitoneal (TEP) hernia repair
  Interventions: Procedure: TEP with fixation
- TAPP without fixation (Experimental): Standard transabdominal preperitoneal (TAPP) hernia repair without mesh fixation
  Interventions: Procedure: TAPP without fixation
- TAPP with fixation (Active Comparator): Standard transabdominal preperitoneal (TAPP) hernia repair
  Interventions: Procedure: TAPP with fixation

INTERVENTIONS:
Procedure: TEP without fixation — Standard totally extraperitoneal preperitoneal (TEP) inguinal hernia repair
  Other Names: TEP no fixation
  Arms: TEP without fixation
Procedure: TEP with fixation — Standard totally extraperitoneal preperitoneal (TEP) inguinal hernia repair
  Other Names: Standard TEP
  Arms: TEP with fixation
Procedure: TAPP without fixation — Standard transabdominal preperitoneal (TAPP) inguinal hernia repair without mesh fixation
  Other Names: TAPP no fixation
  Arms: TAPP without fixation
Procedure: TAPP with fixation — Standard transabdominal preperitoneal (TAPP) inguinal hernia repair
  Other Names: Standard TAPP
  Arms: TAPP with fixation

SUMMARY:
Although mesh fixation has been associated to an increased incidence of nerve injury and involves increased operative costs, many surgeons feel that fixation is necessary to reduce the risk of hernia recurrence. The aim of this study is to evaluate the outcomes of laparoscopic herniorrhaphies performed with and without mesh fixation at our institution.

DETAILED DESCRIPTION:
A randomized prospective study was conducted. Four groups of patients were constituted: (1) TEP with mesh fixation (2) TEP without fixation, (3) TAPP with mesh fixation, (4) TAPP without fixation. 120 patients were randomized to each group. The principal outcomes assessed were postoperative chronic groin pain assessed by visual analogue pain scale (VAS), hernia recurrence, other morbidity rates and hospital costs. Patients were reviewed in outpatient unit at 1 week and at 1, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hernia
* uncomplicated hernia
* medical fitness for general anesthesia

Exclusion Criteria:

* unfit for general anesthesia
* complicated hernia
* uncorrectable coagulopathy
* BMI > 35
* concomitant pathologies requiring simultaneous surgery
* bilateral hernia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-05; Primary Completion 2014-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from preoperative pain levels at 2 years assessed by the visual analogue pain scale (VAS) | preoperative and postoperative 2nd year
  neuralgia, inguinal
Change from preoperative pain levels at 1 year assessed by the VAS | preoperative and postoperative 1st year
  neuralgia, inguinal
Change from preoperative pain levels at 6 months assessed by the VAS | preoperative and postoperative 6th month
  neuralgia, inguinal
Change from preoperative pain levels at 3 months assessed by the VAS | preoperative and postoperative 3th month
  neuralgia, inguinal
Change from preoperative pain levels at 1 month assessed by the VAS | preoperative and postoperative 1 month
  neuralgia, inguinal
Change from preoperative pain levels at 1 week assessed by the VAS | preoperative and postoperative 1th week
  neuralgia, inguinal

SECONDARY OUTCOMES:
Total hospital costs | up to 24 months
  consisted all costs of hospital stays and outpatient treatments
conversion rate | through the first day
  conversion to open surgery
recurrence rate | up to 24 months
  clinical and radiological diagnosed
rate of minor and major complications | 2 year
  it was assessed as; no complication, minor complications, major complications and complications needed reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, M.D., Principal Investigator — Bahçeşehir Üniversitesi Tıp Fakültesi; Onder Ozcan, M.D., Study Chair — Mugla University, School of Medicine
Locations (1):
- Medical Park Gaziantep Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes